CLINICAL TRIAL: NCT01440114
Title: The Effect of Intravenous Fentanyl Prior the End of Surgery on Emergence Agitation in Paediatric Patients After General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Ngamjit Pattaravit, Doctor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PSUEA1
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Agitation
Keywords: emergence agitation; pediatric patient; fentanyl; incidence of emergence agitation; severity of emergence agitation; adverse outcome from intervention
MeSH Terms: conditions — Psychomotor Agitation; Emergence Delirium | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fentanyl group (Active Comparator): First arm: intervention group. Patient in this group received fentanyl 1 mcg/kg (concentration 10mcg/ml) intravenous route 15 minutes before the end of surgery.
  Interventions: Drug: fentanyl
- controlled group (Placebo Comparator): patient in this group received NSS 0.1 ml/kg 15 minutes before the end of surgery
  Interventions: Drug: NSS

INTERVENTIONS:
Drug: fentanyl — In intervention group patient received fentanyl 1 mcg/kg intravenous 15 minutes before the end of surgery.
  Arms: fentanyl group
Drug: NSS — Patient in this group received NSS (0.1ml/kg)intravenous route 15 minutes before the end of surgery.
  Arms: controlled group

SUMMARY:
The propose of this study is to determine the effect of intravenous fentanyl prior the end of surgery on the incidence and severity of EA in pediatric patient.

DETAILED DESCRIPTION:
Emergence agitation (EA) is a common self limiting problem after emerging from general anesthesia (GA) especially in pediatric patients. The incidence of EA in Thai population, the incidences of EA 43.2% in pediatric patients aged between 2-9 years. There have been many studies tried to reduce the incidence of EA in various ways such as Preoperative anxiety reduction method and medication. Premedication, Sedative drugs and narcotic drugs were used to reduce the incidence of EA.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 2-9 years
* IPD patient
* Receiving Chloral hydrate 50mg/kg (BW<20 kgs)or midazolam 0.1 mg /kg (BW>20 kgs)Per oral for premedication
* Scheduled for one kind of these surgeries; Otolaryngology, Ophthalmology, Urology, Orthopedic,General surgery, Plastic surgery and Cardiac catheterization.

Exclusion Criteria:

* ASA physical status IV-V
* History of drug allergy:thiopental, fentanyl cisatracurium, chloral hydrate and diazepam

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
the incidence of emergence agitation | pt was observed since emerging from anesthesia up to 60 minutes

SECONDARY OUTCOMES:
severity of emergence agitation | pt was observed since emerging from anesthesia up to 60 minutes
adverse effect from intravenous fentanyl prior the end of surgery | pt was observed since emerging from anesthesia upto 60 minutes
post operative pain | pt was observed since emerging from anesthesia up to 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand